CLINICAL TRIAL: NCT01730404
Title: A Randomised, Double-blind, Double-dummy, Placebo and Active-controlled, Three-way Crossover Study to Evaluate the Safety, Tolerability and Efficacy of 28-day Inhaled CHF 6001 DPI (1200 µg Daily) in Subjects With COPD
Brief Title: Safety, Tolerability and Efficacy of 28-day Inhaled CHF 6001 DPI in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1201-PR-0079
Record Dates: First submitted 2012-08-23; First posted 2012-11-21 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF6001 (Experimental): CHF6001 DPI (Dry Powder Inhaler) once daily
  Interventions: Drug: CHF6001 DPI
- Roflumilast (Active Comparator): Roflumilast, tablet, once daily
  Interventions: Drug: Roflumilast
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF6001 DPI
  Arms: CHF6001
Drug: Roflumilast
  Arms: Roflumilast
Drug: Placebo
  Arms: placebo

SUMMARY:
Phase IIa study in COPD patients aimed to evaluate the safety, tolerability ,pharmacodynamics (effect on biological markers of inflammation in induced sputum and in blood, and on pulmonary function) and on pharmacokinetics of CHF 6001 (a PDE4 inhibitor) after 28-days of daily inhaled dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures.
2. Male or female aged between 40 and 70 years inclusive.
3. Current or past smoker of at least 10 pack/years
4. BMI in the range of 18-35 Kg/m2
5. GOLD Stage 2 and 3 COPD subjects
6. A history of chronic bronchitis defined as chronic cough and sputum production
7. At screening, subjects must be able to produce an adequate induced sputum sample
8. Female subjects: post-menopausal women having at least 12 months of natural (spontaneous) amenorrhea, or women of childbearing potential using two acceptable methods of contraception for the duration of the study and for the following three months

Exclusion criteria:

1. Female subjects: pregnant or lactating women
2. Past or current history of asthma
3. History of clinically significant hypotensive episodes
4. History or symptoms of significant cardiovascular disease
5. History or symptoms of significant neurological disease
6. Unstable concurrent disease
7. An abnormal and clinically significant 12-lead ECG
8. Clinically relevant abnormal laboratory values
9. Use of oral or systemic corticosteroids oral and/or nebulised Beta2 agonists and/or antibiotics within 6 weeks preceding the screening visit
10. Moderate or severe hepatic impairment (Child-Pugh B or C)
11. Intolerance/hypersensitivity or any contraindication to treatment with roflumilast, tiotropium bromide or salbutamol or any of the excipients contained in the formulations used in the study
12. Chronic use of any other medication for treatment of lung disease like xanthines, antileukotrienes, systemic and inhaled corticosteroids, long acting beta2- agonists, roflumilast (other than the study drug) and cromoglycates
13. Long term (at least 12 hours daily) use of oxygen therapy for chronic hypoxemia.
14. Having received an investigational medicinal drug within 30 days prior to study entry
15. Blood draws of 250 mL or more within 45 days prior to enrolment into the study.
16. Known respiratory disorders other than COPD.
17. History of alcohol dependency, or substance abuse
18. Inability to comply with the study Protocol for any other reason.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adverse events, adverse drug reactions, serious adverse. | After 28 days of treatment
  The number and percentage of subjects experiencing AEs, ADRs, serious AEs and AEs leading to study withdrawal.
Vital signs | After 28 days of treatment
12-lead ECG parameters | After 28 days of treatment

SECONDARY OUTCOMES:
Pharmacokinetics of CHF 6001 and its metabolites | After 28 days of treatment
Induction of sputum | After 28 days of treatment
  Biomarkers of inflammation
Baseline Dyspnea Index and Transition Dyspnea Index Questionnaire | After 28 days of treatment
Lung function measurements | After 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit Ltd; Anthony DeSoyza, MD, Principal Investigator — Freeman Health System; Stephen Smith, MD, Principal Investigator — Celerion; Tim Harrison, MD, Principal Investigator — Nottingham University Hospitals NHS Trust; Muna Albayaty, MD, Principal Investigator — Parexel, early phases
Locations (5):
- Celerion, Belfast, Ireland
- United Kingdom (4):
  - Parexel, early phases, Harrow
  - Medicines Evaluation Unit Ltd, Manchester
  - Freeman Hospital, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2012-001005-25